CLINICAL TRIAL: NCT03200665
Title: Sonographic Evaluation of Fetal Growth in the Third Trimester of Low-risk Pregnancy: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Santa Maria, Portugal (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Catarina Policiano, Principal Investigator, Hospital de Santa Maria, Portugal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FCTUltrasoundIUGR
Record Dates: First submitted 2017-06-24; First posted 2017-06-27 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Condition of Fetal Growth or Malnutrition (Diagnosis)
MeSH Terms: conditions — Malnutrition; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound 35-36 (6 / 7 days weeks) (Experimental): The patients that are randomized to this group, besides accomplishing the standard of care of national guidelines (third trimester ultrasound at 30-32 (6 / 7 days weeks)) will be submitted to an additional third trimester ultrasound at 35-36 (6 / 7 days weeks).
  Interventions: Diagnostic Test: Ultrasound 35-36 (6 / 7 days weeks)
- Standard of Care (No Intervention): This is the control group that will be managed in accordance to national guidelines of screening of late fetal growth restriction in low risk pregnancies: third trimester ultrasound at 30-32 (6 / 7 days weeks).

INTERVENTIONS:
Diagnostic Test: Ultrasound 35-36 (6 / 7 days weeks) — An obstetric ultrasound will be performed at 35-36 (6 / 7 days weeks) including biometric parameters and functional parameters of the fetus
  Arms: Ultrasound 35-36 (6 / 7 days weeks)

SUMMARY:
Sonographic fetal weight estimation at the last weeks of third trimester in low-risk pregnancies is an effective method for diagnosis of fetal growth restriction (FGR) permitting close surveillance and timely delivery. The need for a systematic ultrasound evaluation at the last weeks of a low-risk pregnancy and the best time to perform it remains controversial. The most commonly used clinical screening tool in this population is the serial measurement of symphysis-fundus distance, which is a method of a variable and low sensitivity for detection of FGR.

In Portugal, in accordance with guidelines of Direcção Geral de Saúde from 2015, fetal growth restriction screening in low risk pregnancies is performed with an ultrasound for fetal weight estimation at 30th-33rd weeks. Nonetheless, recent data from randomized trials showed that FGR detection rate was superior at 36 vs 32 weeks' gestation. In cases of severe FGR, detection rate was also superior at 36 vs 32 weeks' gestation. In a prior retrospective study, our group analyzed 1429 term low risk pregnancies and the investigators concluded that small for gestational age term babies (birthweight < 10th centile) had a statistically significant higher rate of operative deliveries for intrapartum fetal distress than appropriate for gestational age as well as a higher rate of admission to neonatal intensive care unit. Moreover the investigators compared the same outcomes within small for gestational age neonates with antepartum detection at 30th-33rd weeks ultrasound vs undetected (normal 30th-33rd weeks ultrasound). Antepartum detection of small for gestational age neonates showed a statistically significant lower rate of operative deliveries for intrapartum fetal distress than undetected small for gestational age neonates. The investigators will conduct a prospective randomized clinical trial with the aim to evaluate if a 35th-37th weeks after the standard of care ultrasound in low risk pregnancies is effective in improving the detection rate of FGR and in reducing cesarean deliveries for intrapartum fetal distress and admission to neonatal intensive care unit.

DETAILED DESCRIPTION:
The population to include in this study corresponds to the low-risk pregnant women with surveillance at the Prenatal Consultation or referenced by the Primary Care units to the Department of Obstetrics & Gynecology of Hospital de Santa Maria. The screening method for detection of fetuses at risk of fetal growth restriction currently used in low-risk pregnancies is the measurement of the symphysis-uterine distal distance at all visits from 24 weeks and a third trimester ultrasound at 30-32 (6 / 7 days weeks).

The patients who agree to participate in the study, after signing an informed consent, will be randomized into 2 groups (with and without an additional ultrasound evaluation at 35-35+6 (6 / 7 days weeks)). The randomization will be done through computer software.

Clinical data will be recorded such as: maternal age, ethnicity, parity, height, weight, socioeconomic status and smoking habits.

In the study group (ultrasound evaluation at 35-35+6 (6 / 7 days weeks)), the ultrasound evaluation will include biometric parameters of the fetus: cephalic perimeter, biparietal diameter, abdominal circumference and femur length. Based on these measurements, the computer system (Astraia) provides the estimated fetal weight and respective percentile according to the Hadlock formula. Amniotic fluid will also be measured (maximum column). Functional evaluation will include: Doppler of the umbilical artery, middle cerebral artery and Uterine arteries. The respective index of pulsatility and cerebroplacental ratio will be registered. All Doppler evaluations will be performed in the absence of somatic and respiratory fetal movements, under transitory maternal apnea, with the lowest insonation angle possible and at least 3 successive complexes will be evaluated for each measurement.

Obstetric and neonatal outcomes will be registered after delivery by revising medical records such as: gestational age at delivery, prepartum hemoglobin, type of labor (spontaneous or induced and respective indication), type of delivery (eutocic, instrumental, antepartum or intrapartum cesarean section), indication of instrumental or cesarean delivery, cardiotocographic register characteristics (repeated severe variable decelerations, late decelerations, absence of variability), evidence of meconial fluid, neonatal morbidity (hypoglycemia, hypothermia, transient tachypnea, hyperbilirubinemia requiring phototherapy, meconium aspiration syndrome, admission to neonatal intensive care unit, metabolic acidosis, intraventricular hemorrhage, necrotizing enterocolitis, sepsis, seizures and asphyxia) and mortality.

Sample size calculation

According to a retrospective analysis performed in the target population of this study, the rate of intrapartum fetal hypoxia requiring obstetric intervention in pregnant women with fetal growth restriction is 28%. Aiming to reduce this adverse perinatal outcome by 10%, it is estimated that the investigators will need to include a total sample of 2700 pregnant women (1350 in each group), with 80% power and α level of 0.05.

Performing third-trimester ultrasound at 30-32 weeks, the rate of antenatal detection of fetal growth restriction is 20.5% in low risk pregnancies. Aiming to increase the detection rate by at least 7%, the investigators will require a total sample of 1,200 pregnant women (600 in each group), with 80% power and α level of 0.05. Thus an interim analysis is expected to be performed when 1200 cases are recruited to the study to compare the detection rate of fetal growth restriction between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Single fetus pregnancy

Exclusion Criteria:

* Diabetes
* Hypertension
* Pre-eclampsia
* Autoimmune diseases
* Antecedent of fetal growth restriction or pre-eclampsia
* Placental anomalies
* Fetal malformations
* Chromosome anomalies
* TORCH Infections

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Patient eligibility is based on gender identity because we will include only pregnant women
Enrollment: 1093 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
To increase the detection rate of late fetal growth restriction in low risk pregnancies | It will be assessed when the baby is delivered (about 5 weeks after intervention) by comparing antenatal fetal weight estimation centiles of both ultrasounds with birthweight centiles and evaluate which ultrasound is more accurate
  Diagnosis of fetal growth restriction is defined as birthweight under 10th centile according to gestational age

SECONDARY OUTCOMES:
To decrease the rate of cesarean and instrumental deliveries indicated by intrapartum hypoxia | It will be assessed after delivery (about 5 weeks after intervention)
  Intrapartum hypoxia will be defined by interpreting continuous cardiotocographic monitoring during labor.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Policiano, Principal Investigator — CHLN, Hospital de Santa Maria. Faculdade de Medicina da Universidade de Lisboa
Locations (1):
- CHLN, Hospital de Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided